CLINICAL TRIAL: NCT01878747
Title: Healthcare Provider Behavior and Children's Perioperative Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Zeev Kain, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCIANES02
Record Dates: First submitted 2013-02-08; First posted 2013-06-17 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative; Infant Behavior
Keywords: Pediatric; Pain; Postoperative; General Anesthesia; Anesthesia Recovery Period; Infant Behavior; Adolescent Behavior; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Infant Behavior; Pain; Adolescent Behavior; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P-TIPS group (Experimental): Provider Tailored Intervention for Perioperative Stress (P-TIPS) aims at reducing preoperative anxiety in children via modifying adults' behavior.P-TIPS program is developed from the proximal-distal theory that suggested that in acute procedural settings specific adult behaviors directly affect children's distress and coping behaviors.
  Interventions: Behavioral: Provider Tailored Intervention for Perioperative Stress
- Control Group (No Intervention): Subjects in this group will not be trained with the P-TIPS method. They will receive a 2-hour seminar on the management of preoperative anxiety and postoperative pain and otherwise will provide standard care to patients.

INTERVENTIONS:
Behavioral: Provider Tailored Intervention for Perioperative Stress — Provider Tailored Intervention for Perioperative Stress (P-TIPS) is developed based on the proximal-distal theory that suggested that in acute procedural settings specific adult behaviors directly affect children's distress and coping behaviors. P-TIPS aims at reducing preoperative anxiety in children via modifying adults' behavior.
  Other Names: P-TIPS
  Arms: P-TIPS group

SUMMARY:
The goal of this randomized trial is to examine the effectiveness of a Provider Tailored Intervention for Perioperative Stress (P-TIPS) in preventing high anxiety and improving the recovery process in children undergoing surgery. Four hospitals and all Healthcare Providers (HCP) in it will be randomized to either a P-TIPS Group, who will receive the newly developed intervention, or a Control Group who will receive a 2-hour seminar on the management of preoperative anxiety and postoperative pain and otherwise will provide standard care. The aims of this study are to:

PRIMARY AIM

1. Determine if P-TIPS is more effective than standard care for preventing high preoperative anxiety among children undergoing anesthesia and surgery. The primary outcome will be observational anxiety in the operating room settings as measured by m-YPAS (modified-Yale Preoperative Anxiety Scale).

SECONDARY AIMS

1. Examine the impact of P-TIPS on surgical recovery parameters such as postoperative pain, recovery room stay, nausea and vomiting, emergence delirium and maladaptive behavioral changes as measured by the PAED, and PHBQ
2. Determine if the use of P-TIPS results in higher satisfaction and lower anxiety scores in the parents.as measured by the STAIs, STAIt and Parent Satisfaction questionnaires
3. Determine if HCP in P-TIPS group display more desired behaviors and less undesired behaviors as compared to control group and whether these behaviors mediate the child and parent-level outcomes.These behaviors will be measured using the m-PCAMPIS

DETAILED DESCRIPTION:
The proposed clustered randomized trial of four children's hospitals: CHOC Children's (CHOC), Children's Hospital Los Angeles (CHLA), Lucile Packard Children's Hospital at Stanford, The Children's Hospital, Denver. At each hospital approximately 20 anesthesia and nursing health care providers (HCP) will examine the effectiveness of a Provider Tailored Intervention for Perioperative Stress (P-TIPS) aimed at preventing high anxiety and improving the recovery process in children undergoing surgery via modifying adults' behavior. Each hospital and all HCP in it will be randomized to either a P-TIPS Group, who will receive the newly developed intervention, or a Control Group who will receive a 2-hour seminar on the management of preoperative anxiety and postoperative pain and otherwise will provide standard care. Objective measures of children's preoperative anxiety and postoperative recovery, as well as adherence measures of HCP will be collected prior and during the experimental period.

HCP in the Intervention group will learn that the use of behaviors as such distraction and medical reinterpretation directs the child's attention towards more enjoyable topics or reframes the procedure into something less threatening, which in turn diverts the child's attention away from their own distress or fear. Conversely, although HCPs often use reassurance and empathy to help soothe children, the education that HCPs receive from P-TIPS will explain that these emotion-focused comments seem to direct children's attention to their own distress and frightening aspects of the medical procedure. HCPs will also learn the intricacies of implementing these strategies and ways to adjust their behavior to effectively keep children engaged in coping related behaviors.

Child's anxiety m-YPAS during induction is assessed at two points, a) entering the operating room and b) introduction of the anesthesia mask to the child. Once in the OR, the child's blood pressure and heart rate is also assessed. A total of 10 child-parent dyad interactions per HCP are collected for the baseline assessment phase. HCP behavior during induction is also videotaped by research assistants and coded later using the P-CAMPIS measure. Also, parents and children answer baseline questionnaires aimed at capturing demographics, anxiety, health beliefs. Postoperative analgesic consumption, behavioral and recovery measures are also collected.

ELIGIBILITY:
INCLUSION CRITERIA:

Children:

* Children who are scheduled to undergo outpatient T&A
* Children whose health status is American Society of Anesthesiologists (ASA) physical status I-III will be recruited for this study
* Only children who are in the normal range of development will be recruited for this study

Parents: Parents of children who are enrolled in the study.

Healthcare Provider:

* Anesthesia care providers in the four study hospitals
* Nurses who provide preoperative nursing care to children who are about to undergo surgery in the four study hospitals

EXCLUSION CRITERIA

Children:

* Patients with health status defined by ASA status IV-V
* Patients who are taking psychotropic medications that affect emotion modulation
* Patients who are taking medications such as erythromycin that interfere with the metabolism of midazolam
* Patients born before 36 weeks gestational age are considered premature and will not be included in this study
* Patients with a positive sleep study and patients who have any indication to be admitted postoperatively (e.g. positive sleep study)
* Patients with a positive sleep study indicating sleep apnea will also be excluded from this study.

Parents:

* Parents who refuse to be part of the study
* Parents who don't speak English if the health care providers involved with that child-parent dyad don't speak the language that is spoken by the parent and child

Healthcare Providers:

* Anesthesiologists who refuse to be part of the study
* Nurses who refuse to be part of the study

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1471 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Child's anxiety in the operating room settings. | 1 day
  m-YPAS (modified-Yale Preoperative Anxiety Scale)

SECONDARY OUTCOMES:
Impact of the intervention on the child's recovery parameters including emergence delirium, systolic pressure, diastolic pressure, heart rate recordings, and analgesic consumption. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zeev N. Kain, MD, MBA, Principal Investigator — UC Irvine Medical Center, Dept. of Anesthesiology and Perioperative Care
Locations (6):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Menlo Park, California
  - CHOC Children's Hospital, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Boyd Graduate Studies Research Center, Athens, Georgia
- IWK Health Center, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Stevenson RS, Rosales A, Fortier MA, Campos B, Golianu B, Zuk J, Gold J, Kain ZN. The Role of Ethnicity and Acculturation in Preoperative Distress in Parents of Children Undergoing Surgery. J Immigr Minor Health. 2017 Jun;19(3):738-744. doi: 10.1007/s10903-016-0357-7. PMID 26895152